CLINICAL TRIAL: NCT06952283
Title: Effects of Music Intervention on Golf-Specific Skill Performance of Chinese Golfers Under Mental Fatigue
Brief Title: Music Intervention on Golfers Under Mental Fatigue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pan Xiaoyang (Other)
Responsible Party: Sponsor-Investigator, Pan Xiaoyang, PhD Candidate, Department of Sport Studies, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUSOM2025-066
Record Dates: First submitted 2025-04-09; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Mental Fatigue
Keywords: lack of energy; feelings of tiredness; decreased attention; impaired cognitive; impaired behavioral performance
MeSH Terms: conditions — Mental Fatigue; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization of group allocation and participant order will be conducted using a random number table generator (www.randomizer.org), ensuring that no one can predict the group assignments before randomization. Participants will not be informed of the true purpose of the study; instead, they will be told that the study is part of a quarterly training program and that they should perform their best during the skill testing phase. During the intervention, dedicated assistants will be responsible for inducing mental fatigue and administering the music intervention, but they will not be informed of the specific research objectives. During the golf skill testing and performance recording phase, testing assistants will be responsible only for recording test results and will not be aware of the participants' group assignments. Data analysis will be conducted by researchers who only have access to anonymized data, further reinforcing blinding control. Group assignment information will only be
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MF-Mu Group (Experimental): MF-Mu Group: Participants undergo a mental fatigue induction task followed by a music intervention
  Interventions: Behavioral: Inducing mental fatigue; Behavioral: Music intervention
- MF-nMu Group (Active Comparator): MF-nMu Group: Participants undergo a mental fatigue induction task but do not receive a music intervention
  Interventions: Behavioral: Inducing mental fatigue
- CON Group (No Intervention): CON Group: Participants neither undergo a mental fatigue induction task nor receive a music intervention

INTERVENTIONS:
Behavioral: Inducing mental fatigue — During the mental fatigue induction phase, a 30-minute Stroop task will artificially induce mental fatigue, simulating the mental fatigue state that athletes experience during competitions or training sessions. The Stroop task is a classic cognitive control task widely used for inducing mental fatigue. Research in sports science has shown that a 30-minute Stroop task significantly increases subjective fatigue and reduces physical performance. This study will use a smartphone-based version of the Stroop task (with brightness and touch sensitivity standardised), where colour words (such as "red" and "blue") are displayed continuously, but the font colour does not match the word's meaning. Participants must ignore the word's meaning and respond only based on the font colour. The Stroop task requires sustained attention, conflict resolution, and cognitive inhibition, leading to cognitive resource depletion and mental fatigue accumulation.
  Arms: MF-Mu Group; MF-nMu Group
Behavioral: Music intervention — During the music intervention phase, participants will listen to 15 minutes of classical music to facilitate mental fatigue recovery. This study selects Mozart's Eine Kleine Nachtmusik as the intervention music, a piece that has been applied in previous mental fatigue recovery studies and has been validated as an effective intervention. The intervention duration is set at 15 minutes, as multiple studies have confirmed this duration to be sufficient to produce recovery effects without causing additional cognitive load or auditory fatigue. The music will be played through a smartphone, with the intervention volume controlled at 50-60 dBA. Considering that the maximum volume of a smartphone is approximately 105-113 dBA, the standardised intervention volume is set at 50% (52.5-56.5 dBA) of the smartphone's maximum volume to ensure consistency among all participants.
  Arms: MF-Mu Group

SUMMARY:
This study aims to evaluate the effects of music intervention on golf-specific skill performance under mental fatigue. It is a randomised, controlled, double-blind design. The study consists of three main phases: familiarisation with the experimental procedure, baseline testing, and the formal experiment. During the formal experiment, participants will be randomly assigned to one of the following three groups: (MF-Mu Group) Participants undergo a mental fatigue induction task followed by a music intervention; (MF-nMu Group) Participants undergo a mental fatigue induction task but do not receive a music intervention; (CON Group) Participants neither undergo a mental fatigue induction task nor receive a music intervention. The total intervention duration is 45 minutes, consisting of 30 minutes of mental fatigue induction and 15 minutes of music intervention. In conditions where mental fatigue induction or music intervention is not conducted, participants will remain in the same experimental environment and rest quietly for the same duration to control for external confounding factors and ensure experimental consistency. Immediately after the intervention, participants will complete golf skill testing, with the testing site located within a 2 minutes walking distance from the intervention area. Performance outcomes include driving performance, iron shot performance, chipping performance, and putting performance.

ELIGIBILITY:
Inclusion Criteria:

* Athletes must be between 18 and 24 years old.
* Be registered golfers in the National Colleges and Universities Golf Championship.
* Have at least three years of specialised golf training.
* Engage in at least five weekly training sessions.

Exclusion Criteria:

* Colour blindness.
* Hearing loss.
* Insomnia.
* Physical injuries.
* Ongoing mental health issues.
* The use of any medication that might influence cognitive.
* The use of any medication that might influence physical performance.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The change in golf driving accuracy after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The golf driving performance test follows the Golf Skill Level Standards and Testing Methods issued by the China Golf Association, assessing accuracy. The target is located 210 yards from the hitting area, and expands outward at an angle, widening to approximately 20 yards additional space on either side. Accuracy is determined by the number of balls landing in the designated target area. A total of 10 shots are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
The change in golf driving shot quality after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The driving shot quality is evaluated based on the golfer's subjective feedback after each shot, responding to the question: "Do you think this shot was solid?" Responses are recorded as "Yes" (solid contact) or "No" (poor contact). A total of 10 shots are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
The change in iron shot accuracy after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (after the driving test) (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The 150 yards iron shot performance test follows the Golf Skill Level Standards and Testing Methods issued by the China Golf Association, assessing accuracy. The distance to the target is 150 yards. The Target Zone is a rectangle positioned 150 yards away, measuring 20 yards wide and 30 yards deep (15 yards before and 15 yards after the 150-yard line). Accuracy is determined by the number of balls landing in the designated target area. A total of 10 shots are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
The change in iron shot shot quality after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (after the driving test) (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The iron shot quality is evaluated based on the golfer's subjective feedback after each shot, responding to the question: "Do you think this shot was solid?" Responses are recorded as "Yes" (solid contact) or "No" (poor contact). A total of 10 shots are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
The change in chipping accuracy after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (after the iron test) (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The 30 yards chipping performance test follows the Golf Skill Level Standards and Testing Methods issued by the China Golf Association, assessing accuracy. The distance to the target is 30 yards. The Target Zone is a circular area with a 3-yard radius around the hole. Accuracy is determined by the number of balls landing in the designated target area. A total of 10 shots are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
The change in chipping shot quality after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (after the iron test) (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The chipping shot quality is evaluated based on the golfer's subjective feedback after each shot, responding to the question: "Do you think this shot was solid?" Responses are recorded as "Yes" (solid contact) or "No" (poor contact). A total of 10 shots are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
The change in putting accuracy after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (after the chipping test) (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The putting performance test follows the Golf Skill Level Standards and Testing Methods issued by the China Golf Association, assessing accuracy . Participants perform putts of two different distances from the Ball-striking Zone. A successful putt is defined as either holing the ball (for the 1.5-yard putt) or stopping the ball within the 1-yard radius Target Zone (for the 7-yard putt). A total of 10 shots (5 1.5-yard putt and 5 7-yard putt) are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
The change in putting shot quality after music intervention compared to performance under mental fatigue. | Baseline and immediately after the music intervention (after the chipping test) (No more than 40 seconds per shot, with a total duration of about 5 minutes).
  The putting shot quality is evaluated based on the golfer's subjective feedback after each shot, responding to the question: "Do you think this shot was solid?" Responses are recorded as "Yes" (solid contact) or "No" (poor contact). A total of 10 shots are performed, with 1 point awarded per successful shot, resulting in a score range of 1 to 10 points.
Mental fatigue | Baseline, before mental fatigue induction, immediately after mental fatigue induction, and immediately after the music intervention (about 30 seconds per test).
  The Visual Analog Scale (VAS) assesses participants' subjective perception of mental fatigue. The scoring is based on a 100 mm linear scale, where participants mark a point between 0 (none at all) and 100 (extremely intense) to describe their current level of mental fatigue.

SECONDARY OUTCOMES:
Immersive Tendency | Baseline (about 1 minute).
  The Immersive Tendency Questionnaire (ITQ) assesses participants' degree of immersion in the virtual environment (music). This questionnaire consists of 18 items categorised into four factors: immersive tendency, individual alertness, physical state, and attention-shifting ability. Each item is rated on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Motivation | Baseline, before mental fatigue induction, immediately after mental fatigue induction, and immediately after the music intervention (about 30 seconds per test).
  The Visual Analog Scale (VAS) assesses participants' subjective perception of motivation levels. The scoring is based on a 100 mm linear scale, where participants mark a point between 0 (none at all) and 100 (extremely intense) to describe their current level of motivation.
Sport Anxiety | Baseline, before mental fatigue induction, immediately after mental fatigue induction, and immediately after the music intervention (about 1 minute per test).
  The Sport Anxiety Scale-2 (SAS-2) assesses participants' trait sport anxiety levels. This scale consists of 15 items categorised into three factors: somatic anxiety, worry, and concentration disruption. Each item is rated on a 4-point Likert scale, ranging from 1 (not at all) to 4 (very much so).
Rating Perception of Effort | Baseline, before mental fatigue induction, immediately after mental fatigue induction, and immediately after the music intervention (about 30 seconds per test).
  The Borg Rating of Perceived Exertion (Borg RPE) assesses individuals' subjective effort levels. This scale employs a 15-level scoring system, ranging from 6 (extremely easy) to 20 (extremely strenuous), to reflect athletes' subjective perception of workload intensity during testing or competition.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Geok Soh, Prof. Dr., Study Director — Department of Sport Studies, Faculty of Educational Studies, Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share IPD, although this may be reconsidered in the future depending on data privacy safeguards, participant consent, and availability of secure sharing platforms.

REFERENCES:
- [Background] Abbasi M, Esmaeili R, Pourabdian S, Shakerian M. Exploring the influence of music on cognitive performance in female assembly line workers at a medical device manufacturing unit. PLoS One. 2024 Oct 23;19(10):e0309555. doi: 10.1371/journal.pone.0309555. eCollection 2024. PMID 39441850
- [Background] Arenales Arauz YL, Habay J, Ocvirk T, Mali A, Russell S, Marusic U, De Pauw K, Roelands B. The interplay of brain neurotransmission and mental fatigue: A research protocol. PLoS One. 2024 Sep 10;19(9):e0310271. doi: 10.1371/journal.pone.0310271. eCollection 2024. PMID 39255295
- [Background] Axelsen JL, Kirk U, Staiano W. On-the-spot binaural beats and mindfulness reduces the effect of mental fatigue. Journal of Cognitive Enhancement. 2020 Mar;4(1):31-9. https://doi.org/10.1007/s41465-019-00162-3
- [Background] Azevedo R, Silva-Cavalcante MD, Gualano B, Lima-Silva AE, Bertuzzi R. Effects of caffeine ingestion on endurance performance in mentally fatigued individuals. Eur J Appl Physiol. 2016 Dec;116(11-12):2293-2303. doi: 10.1007/s00421-016-3483-y. Epub 2016 Sep 30. PMID 27695980
- [Background] Bhandarkar S, Salvi BV, Shende P. Current scenario and potential of music therapy in the management of diseases. Behav Brain Res. 2024 Feb 26;458:114750. doi: 10.1016/j.bbr.2023.114750. Epub 2023 Nov 8. PMID 37944563
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Cao S, Geok SK, Roslan S, Sun H, Lam SK, Qian S. Mental Fatigue and Basketball Performance: A Systematic Review. Front Psychol. 2022 Jan 10;12:819081. doi: 10.3389/fpsyg.2021.819081. eCollection 2021. PMID 35082736
- [Background] Caparros-Gonzalez RA, de la Torre-Luque A, Diaz-Piedra C, Vico FJ, Buela-Casal G. Listening to Relaxing Music Improves Physiological Responses in Premature Infants: A Randomized Controlled Trial. Adv Neonatal Care. 2018 Feb;18(1):58-69. doi: 10.1097/ANC.0000000000000448. PMID 29045255
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Colin C, Prince V, Bensoussan JL, Picot MC. Music therapy for health workers to reduce stress, mental workload and anxiety: a systematic review. J Public Health (Oxf). 2023 Aug 28;45(3):e532-e541. doi: 10.1093/pubmed/fdad059. PMID 37147921
- [Background] Cosmo BG, de Menezes Vervloet G, Rocha JP, Klein MP, dos Santos Silva R, Campos VR. Music therapy as a non-pharmacological intervention in Alzheimer's disease: an integrative review. Rev Med (São Paulo). 2022 Sep;101(5):197832. https://doi.org/10.11606/issn.1679-9836.v101i5e-197832
- [Background] Ding C, Kim Geok S, Sun H, Roslan S, Cao S, Zhao Y. Does music counteract mental fatigue? A systematic review. PLoS One. 2025 Jan 3;20(1):e0316252. doi: 10.1371/journal.pone.0316252. eCollection 2025. PMID 39752412
- [Background] Du YJ, Guan YH, Thome KT, Dong JC. Music Therapy and Music Intervention for NSCLC Patients Undergoing PET with Fear of Cancer Recurrence. Integr Cancer Ther. 2024 Jan-Dec;23:15347354241269898. doi: 10.1177/15347354241269898. PMID 39135426
- [Background] Englert C, Bertrams AG. Active relaxation counteracts the effects of ego depletion on performance under evaluative pressure in a state of ego depletion. Sportwissenschaft. 2016;46(2):110-5. https://doi.org/110-115. 10.1007/s12662-015-0383-y
- [Background] Faro H, Fortes LD, Lima-Junior DD, Barbosa BT, Ferreira ME, Almeida SS. Sport-based video game causes mental fatigue and impairs visuomotor skill in male basketball players. International Journal of Sport and Exercise Psychology. 2023 Nov 2;21(6):1125-39. https://doi.org/10.1080/1612197X.2022.2109187
- [Background] Farrally MR, Cochran AJ, Crews DJ, Hurdzan MJ, Price RJ, Snow JT, Thomas PR. Golf science research at the beginning of the twenty-first century. J Sports Sci. 2003 Sep;21(9):753-65. doi: 10.1080/0264041031000102123. PMID 14579870
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fortes LS, De Lima-Junior D, Fiorese L, Nascimento-Junior JRA, Mortatti AL, Ferreira MEC. The effect of smartphones and playing video games on decision-making in soccer players: A crossover and randomised study. J Sports Sci. 2020 Mar;38(5):552-558. doi: 10.1080/02640414.2020.1715181. Epub 2020 Jan 15. PMID 31941416
- [Background] Fortes LS, Ferreira MEC, Faro H, Penna EM, Almeida SS. Brain Stimulation Over the Motion-Sensitive Midtemporal Area Reduces Deleterious Effects of Mental Fatigue on Perceptual-Cognitive Skills in Basketball Players. J Sport Exerc Psychol. 2022 May 25;44(4):272-285. doi: 10.1123/jsep.2021-0281. Print 2022 Aug 1. PMID 35613846
- [Background] Fortes LS, Lima-Junior D, Barbosa BT, Faro HK, Ferreira ME, Almeida SS. Effect of mental fatigue on decision-making skill and visual search behaviour in basketball players: an experimental and randomised study. International Journal of Sport and Exercise Psychology. 2022 Mar 31:1-20. https://doi.org/10.1080/1612197X.2022.2058055
- [Background] Franco-Alvarenga PE, Brietzke C, Canestri R, Goethel MF, Hettinga F, Santos TM, Pires FO. Caffeine improved cycling trial performance in mentally fatigued cyclists, regardless of alterations in prefrontal cortex activation. Physiol Behav. 2019 May 15;204:41-48. doi: 10.1016/j.physbeh.2019.02.009. Epub 2019 Feb 10. PMID 30742838
- [Background] Ghetti CM. Music therapy as procedural support for invasive medical procedures: Toward the development of music therapy theory. Nordic Journal of Music Therapy. 2012 Feb 1;21(1):3-5. https://doi.org/10.1080/08098131.2011.571278
- [Background] Grafton-Clarke C, Grace L, Harky A. Music therapy following cardiac surgery-is it an effective method to reduce pain and anxiety? Interact Cardiovasc Thorac Surg. 2019 May 1;28(5):722-727. doi: 10.1093/icvts/ivy311. PMID 30508181
- [Background] Guerrero JM, Castano PM, Schmidt EO, Rosario L, Westhoff CL. Music as an auxiliary analgesic during first trimester surgical abortion: a randomized controlled trial. Contraception. 2012 Aug;86(2):157-62. doi: 10.1016/j.contraception.2011.11.017. Epub 2012 Jan 10. PMID 22240180
- [Background] Habay J, Van Cutsem J, Verschueren J, De Bock S, Proost M, De Wachter J, Tassignon B, Meeusen R, Roelands B. Mental Fatigue and Sport-Specific Psychomotor Performance: A Systematic Review. Sports Med. 2021 Jul;51(7):1527-1548. doi: 10.1007/s40279-021-01429-6. Epub 2021 Mar 12. PMID 33710524
- [Background] Han J, Xie H, Cong S, Wang M, Ni S, Wu Y, Zhang A. Effectiveness of smartphone-based music intervention on perinatal depression: protocol for a randomized controlled trial. BMC Psychol. 2024 Nov 7;12(1):633. doi: 10.1186/s40359-024-02141-6. PMID 39511663
- [Background] Jacquet T, Poulin-Charronnat B, Bard P, Perra J, Lepers R. Physical Activity and Music to Counteract Mental Fatigue. Neuroscience. 2021 Dec 1;478:75-88. doi: 10.1016/j.neuroscience.2021.09.019. Epub 2021 Sep 30. PMID 34601062
- [Background] Jensen AR, Rohwer WD Jr. The Stroop color-word test: a review. Acta Psychol (Amst). 1966;25(1):36-93. doi: 10.1016/0001-6918(66)90004-7. No abstract available. PMID 5328883
- [Background] Kim G, Han W. Sound pressure levels generated at risk volume steps of portable listening devices: types of smartphone and genres of music. BMC Public Health. 2018 May 1;18(1):481. doi: 10.1186/s12889-018-5399-4. PMID 29712550
- [Background] Klein MO, Battagello DS, Cardoso AR, Hauser DN, Bittencourt JC, Correa RG. Dopamine: Functions, Signaling, and Association with Neurological Diseases. Cell Mol Neurobiol. 2019 Jan;39(1):31-59. doi: 10.1007/s10571-018-0632-3. Epub 2018 Nov 16. PMID 30446950
- [Background] Loch F, zum Berge AH, Kölling S, Kellmann M. Stress states, mental fatigue, and the concept of mental recovery in sports. InFeelings in Sport 2020 Sep 17 (pp. 235-245). Routledge.
- [Background] Lorek M, Bak D, Kwiecien-Jagus K, Medrzycka-Dabrowska W. The Effect of Music as a Non-Pharmacological Intervention on the Physiological, Psychological, and Social Response of Patients in an Intensive Care Unit. Healthcare (Basel). 2023 Jun 8;11(12):1687. doi: 10.3390/healthcare11121687. PMID 37372805
- [Background] Magee WL. Music therapy with patients in low awareness states: approaches to assessment and treatment in multidisciplinary care. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):522-36. doi: 10.1080/09602010443000461. PMID 16350993
- [Background] Martin K, Meeusen R, Thompson KG, Keegan R, Rattray B. Mental Fatigue Impairs Endurance Performance: A Physiological Explanation. Sports Med. 2018 Sep;48(9):2041-2051. doi: 10.1007/s40279-018-0946-9. PMID 29923147
- [Background] McMorris T. Cognitive Fatigue Effects on Physical Performance: The Role of Interoception. Sports Med. 2020 Oct;50(10):1703-1708. doi: 10.1007/s40279-020-01320-w. PMID 32661840
- [Background] Mizuno K, Tanaka M, Yamaguti K, Kajimoto O, Kuratsune H, Watanabe Y. Mental fatigue caused by prolonged cognitive load associated with sympathetic hyperactivity. Behav Brain Funct. 2011 May 23;7:17. doi: 10.1186/1744-9081-7-17. PMID 21605411
- [Background] Mozart WA, Brainin N, Klier M, Lovett M, Nissel S, Schidlof P, Seifert G, Zepperitz R, Quartet AS. Eine kleine Nachtmusik G dur KV 525 Ein musikalischer Spass KV 522" Dorfmusikanten-Sextett". Deutsche Grammophon; 1982.
- [Background] Pageaux B, Lepers R. The effects of mental fatigue on sport-related performance. Prog Brain Res. 2018;240:291-315. doi: 10.1016/bs.pbr.2018.10.004. Epub 2018 Oct 26. PMID 30390836
- [Background] Pageaux B, Lepers R, Dietz KC, Marcora SM. Response inhibition impairs subsequent self-paced endurance performance. Eur J Appl Physiol. 2014 May;114(5):1095-105. doi: 10.1007/s00421-014-2838-5. Epub 2014 Feb 15. PMID 24531591
- [Background] Pan X, Soh KG, Soh KL. Viable strategies for enhancing performance in ball sports by mitigating mental fatigue: A systematic review. PLoS One. 2024 Nov 8;19(11):e0313105. doi: 10.1371/journal.pone.0313105. eCollection 2024. PMID 39514612
- [Background] Pauwels EK, Volterrani D, Mariani G, Kostkiewics M. Mozart, music and medicine. Med Princ Pract. 2014;23(5):403-12. doi: 10.1159/000364873. Epub 2014 Jul 19. PMID 25060169
- [Background] Proost M, Habay J, De Wachter J, De Pauw K, Rattray B, Meeusen R, Roelands B, Van Cutsem J. How to Tackle Mental Fatigue: A Systematic Review of Potential Countermeasures and Their Underlying Mechanisms. Sports Med. 2022 Sep;52(9):2129-2158. doi: 10.1007/s40279-022-01678-z. Epub 2022 May 11. PMID 35543922
- [Background] Qi P, Ru H, Gao L, Zhang X, Zhou T, Tian Y, Thakor N, Bezerianos A, Li J, Sun Y. Neural mechanisms of mental fatigue revisited: New insights from the brain connectome. Engineering. 2019 Apr 1;5(2):276-86. https://doi.org/10.1016/j.eng.2018.11.025
- [Background] VAN Cutsem J, Roelands B, Pluym B, Tassignon B, Verschueren JO, DE Pauw K, Meeusen R. Can Creatine Combat the Mental Fatigue-associated Decrease in Visuomotor Skills? Med Sci Sports Exerc. 2020 Jan;52(1):120-130. doi: 10.1249/MSS.0000000000002122. PMID 31403610
- [Background] Russell S, Jenkins D, Rynne S, Halson SL, Kelly V. What is mental fatigue in elite sport? Perceptions from athletes and staff. Eur J Sport Sci. 2019 Nov;19(10):1367-1376. doi: 10.1080/17461391.2019.1618397. Epub 2019 May 28. PMID 31081474
- [Background] Smith MR, Thompson C, Marcora SM, Skorski S, Meyer T, Coutts AJ. Mental Fatigue and Soccer: Current Knowledge and Future Directions. Sports Med. 2018 Jul;48(7):1525-1532. doi: 10.1007/s40279-018-0908-2. PMID 29623604
- [Background] Smith RE, Smoll FL, Cumming SP, Grossbard JR. Measurement of multidimensional sport performance anxiety in children and adults: The Sport Anxiety Scale-2. Journal of sport and exercise psychology. 2006 Dec 1;28(4):479-501. https://doi.org/10.1123/jsep.28.4.479
- [Background] Sun H, Soh KG, Roslan S, Wazir MRWN, Soh KL. Does mental fatigue affect skilled performance in athletes? A systematic review. PLoS One. 2021 Oct 14;16(10):e0258307. doi: 10.1371/journal.pone.0258307. eCollection 2021. PMID 34648555
- [Background] Sun H, Soh KG, Mohammadi A, Wang X, Bin Z, Zhao Z. Effects of mental fatigue on technical performance in soccer players: A systematic review with a meta-analysis. Front Public Health. 2022 Jul 22;10:922630. doi: 10.3389/fpubh.2022.922630. eCollection 2022. PMID 35937235
- [Background] Sun H, Soh KG, Roslan S, Wazir MRWN, Mohammadi A, Ding C, Zhao Z. Nature exposure might be the intervention to improve the self-regulation and skilled performance in mentally fatigue athletes: A narrative review and conceptual framework. Front Psychol. 2022 Aug 2;13:941299. doi: 10.3389/fpsyg.2022.941299. eCollection 2022. PMID 35983203
- [Background] Tanaka M, Ishii A, Watanabe Y. Neural effects of mental fatigue caused by continuous attention load: a magnetoencephalography study. Brain Res. 2014 May 2;1561:60-6. doi: 10.1016/j.brainres.2014.03.009. Epub 2014 Mar 16. PMID 24642273
- [Background] Terry PC, Karageorghis CI, Curran ML, Martin OV, Parsons-Smith RL. Effects of music in exercise and sport: A meta-analytic review. Psychol Bull. 2020 Feb;146(2):91-117. doi: 10.1037/bul0000216. Epub 2019 Dec 5. PMID 31804098
- [Background] Thompson CJ, Noon M, Towlson C, Perry J, Coutts AJ, Harper LD, Skorski S, Smith MR, Barrett S, Meyer T. Understanding the presence of mental fatigue in English academy soccer players. J Sports Sci. 2020 Jul;38(13):1524-1530. doi: 10.1080/02640414.2020.1746597. Epub 2020 Mar 25. PMID 32212903
- [Background] Van Cutsem J, De Pauw K, Marcora S, Meeusen R, Roelands B. A caffeine-maltodextrin mouth rinse counters mental fatigue. Psychopharmacology (Berl). 2018 Apr;235(4):947-958. doi: 10.1007/s00213-017-4809-0. Epub 2017 Dec 15. PMID 29247343
- [Background] Van Cutsem J, Marcora S, De Pauw K, Bailey S, Meeusen R, Roelands B. The Effects of Mental Fatigue on Physical Performance: A Systematic Review. Sports Med. 2017 Aug;47(8):1569-1588. doi: 10.1007/s40279-016-0672-0. PMID 28044281
- [Background] Waer FB, Alexe DI, Alexe CI, Eken Ö, Păun LI, Sahli S. Impact of classical music listening on cognitive and functional performances in Middle-aged women. Applied Sciences. 2024 Aug 2;14(15):6779. https://doi.org/10.3390/app14156779
- [Background] Wang Z, Xu W, Zhang C, Zhang C, Liu Y, Chen P, Han G, Wang L. Music boosts the recovery of attention after mental fatigue in healthy young male subjects: A human auditory event-related potential study. Behav Brain Res. 2025 May 8;485:115539. doi: 10.1016/j.bbr.2025.115539. Epub 2025 Mar 13. PMID 40089211
- [Derived] Pan X, Soh KG, Jaafar WMW, Sun H, Zhang G. Effects of music intervention on golf-specific skill performance of golfers under mental fatigue: Protocol for a randomized controlled trial. PLoS One. 2025 Dec 4;20(12):e0337905. doi: 10.1371/journal.pone.0337905. eCollection 2025. PMID 41343510